CLINICAL TRIAL: NCT01921530
Title: Interbody Fusion and Decompression Versus Instrumented Posterolateral Fusion and Decompression for Lumbar Spinal Stenosis With Degenerative Spondylolisthesis
Brief Title: Interbody vs Instrumented Posterolateral Fusion Following Decompression for Lumbar Spinal Stenosis With Degenerative Spondylolisthesis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The London Spine Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103386
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Degenerative Spondylolisthesis; Spinal Stenosis
Keywords: Posterolateral Fusion; Interbody Fusion; Lumbar; Spinal Stenosis; Degenerative Spondylolisthesis
MeSH Terms: conditions — Spinal Stenosis

ARMS (2):
- Interbody Fusion (Active Comparator)
  Interventions: Procedure: Interbody Fusion
- Posterolateral Fusion (Active Comparator)
  Interventions: Procedure: Posterolateral Fusion

INTERVENTIONS:
Procedure: Interbody Fusion — The interbody fusion (IF) procedure requires exposure and removal of the disc, curetting the end plates, inserting a cage filled with bone graft, as well as stabilization with rods and screws.
  Other Names: Posterolateral Interbody Fusion (PLIF); Transforaminal Interbody fusion (TLIF)
  Arms: Interbody Fusion
Procedure: Posterolateral Fusion — In posterolateral fusion stabilization is achieved using pedicle screws joined by rods. The graft used to facilitate fusion is placed between decorticated transverse processes and can be an autograft of iliac bone or local bone, allograft, or a synthetic expander.
  Arms: Posterolateral Fusion

SUMMARY:
Degenerative spondylolisthesis describes the slip of one spinal segment relative to the adjacent segment. It is usually associated with spinal stenosis (which limits one's ability to walk and stand) and is the most common indication for surgery in adults over age 65 years. A variety of surgical techniques are available; the most common are the Posterolateral Instrumented Fusion (PLF), and Interbody Fusion (IF) including Posterolateral Interbody Fusion (PLIF), and Transforaminal Interbody fusion (TLIF). IF uses a cage that is placed within the cleaned out disc space between the vertebral bodies being fused. Although this approach achieves a good fusion rate and deformity correction it is associated with a higher surgical cost and potential intra-operative complication rate. What is more, no consensus exists as to whether IF provides better patient rated functional outcome and quality of life. If the advantages of IF do not translate into superior patient rated outcomes, then the risk-benefit ratio would be tipped in favor of PLF. The purpose of this study is to determine if IF is equivalent to PLF for the treatment of degenerative spondylolisthesis. The investigators will conduct a prospective randomized control trial comparing these two procedures. Our primary outcome measure will be the Oswestry Disability Index, which evaluates spinal pain and function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 50 years or older
2. Grade I or II (less than 50% slip of the cephalad vertebra compared to the caudal vertebra) degenerative spondylolisthesis at one or two contiguous levels between L1 and L5.
3. Lumbar spinal stenosis at the same levels of the degenerative spondylolisthesis producing radiculopathy or neurogenic claudication unresponsive to a minimum of 3 months of non surgical treatment
4. Patients who are medically suitable for surgical management
5. Patients who have consented for surgical treatment
6. Patients able to provide informed consent for the study and complete the questionnaires

Exclusion Criteria:

1. Lytic spondylolisthesis
2. Non degenerative stenosis (example: tumor, trauma, epidural lipomatosis)
3. Severe vertical foraminal stenosis necessitating interbody insertion to re-establish foraminal height
4. Segmental kyphosis at the level of the spondylolisthesis
5. Segmental scoliosis >10 degrees at the level of the spondylolisthesis
6. Rheumatoid arthritis
7. Active infection
8. On long term disability or workers compensation claim
9. Drug or alcohol misuse
10. Lack of permanent home residence
11. Previous surgery at the proposed surgical level
12. Previous fusion in the lumbar spine
13. Contraindication to surgery: medical co morbidities
14. Unable to complete questionnaire (e.g. Dementia)
15. Unable to give voluntary consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2013-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | 1 year post surgery
  The Oswestry Disability Index is an effective method of measuring disability in patients with back and leg pain and is well suited to patients who have had persistent severe disability. It is a commonly utilized, validated, and highly reproducible. The questionnaire can be completed in less than 5 minutes and a large amount of normative data exists.

SECONDARY OUTCOMES:
Oswestry Disability Index | Enrollment, and at 6 weeks, 3 months, 6 months, 2 years, 5 years and post surgery
  The Oswestry Disability Index is an effective method of measuring disability in patients with back and leg pain and is well suited to patients who have had persistent severe disability. It is a commonly utilized, validated, and highly reproducible. The questionnaire can be completed in less than 5 minutes and a large amount of normative data exists.

OTHER OUTCOMES:
Visual Analogue Scale for back pain intensity (0-10: 0= no pain, 10=worst pain) | Enrollment at 6 weeks, 3 months, 6 months, 1 year, 2 year, 5 year post surgery
Visual Analogue Scale for leg pain intensity (0-10: 0= no pain, 10=worst pain) | Enrollment and at 6 weeks, 3 months, 6 months, 1 year, 2 year, 5 year post surgery
SF-12 (General Health outcome measure) | Enrollment at 6 weeks, 3 months, 6 months, 1 year, 2 year, 5 year post surgery
  The SF-12 is a standardized health related quality of life outcome questionnaire, which assess 8 health domains. The physical and mental component can be derived. It has been shown to be valid and reliable when applied to the spine patient population.
Patient satisfaction | Enrollment and at 6 weeks, 3 months, 6 months, 1 year, 2 year, 5 year post surgery
  "All things considered, how satisfied are you with the results of your recent treatment for your spine fracture? 1-7, 8= not sure." This sentence is the recommended tool for assessing global satisfaction.
Cost analysis | Enrollment, and at 6 weeks, 3 months, 6 months, 1 year, 2 year, 5 year post surgery
  Prolo economic score and cost analysis for each procedure
Fusion rates | 6 months, 1 year, 5 year
Intra-operative Complication rate | within 6 weeks after sugery

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Bailey, MD, Principal Investigator — The London Spine Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada